CLINICAL TRIAL: NCT01584440
Title: A Phase 2, Randomized, Double-dummy, Double-blind, Placebo-controlled Study to Assess the Efficacy, Safety and Tolerability of AVP-923 (Dextromethorphan/Quinidine) for the Treatment of Symptoms of Agitation in Patients With Alzheimer's Disease.
Brief Title: Efficacy, Safety and Tolerability Study of AVP-923 (Dextromethorphan/Quinidine) for Treatment of Symptoms of Agitation in Participants With Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Avanir Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12-AVR-131
Record Dates: First submitted 2012-04-23; First posted 2012-04-25 (Estimated); Results first posted 2021-11-26 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-10

CONDITIONS: Agitation; Alzheimer's Disease
Keywords: AVP-923-20; AVP-923-30; AVP-923; Dextromethorphan; Quinidine; Neuropsychiatric Inventory; Aggression; Efficacy; Safety
MeSH Terms: conditions — Psychomotor Agitation; Alzheimer Disease; Aggression | interventions — dextromethorphan - quinidine combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Participants will receive placebo during Stage 1 and Stage 2 of the study.
  Interventions: Drug: Placebo
- AVP-923 (Experimental): Participants will receive AVP-923-20 and AVP-923-30 in a sequential manner during Stage 1 and Stage 2 of the study.
  Interventions: Drug: AVP-923-20; Drug: AVP-923-30
- Placebo then AVP-923 (Experimental): Participants will receive placebo in Stage 1 followed by AVP-923 in Stage 2.
  Interventions: Drug: AVP-923-20; Drug: Placebo; Drug: AVP-923-30

INTERVENTIONS:
Drug: AVP-923-20 — AVP-923-20: 20 mg of dextromethorphan and 10 mg of quinidine
  Other Names: Nuedexta
  Arms: AVP-923; Placebo then AVP-923
Drug: Placebo — Placebo capsule
  Arms: Placebo; Placebo then AVP-923
Drug: AVP-923-30 — AVP-923-30: 30 mg of dextromethorphan and 10 mg of quinidine
  Arms: AVP-923; Placebo then AVP-923

SUMMARY:
The objectives of the study are to evaluate the safety, tolerability and efficacy of AVP-923 compared to placebo, for the treatment of symptoms of agitation in participants with Alzheimer's Disease (AD).

DETAILED DESCRIPTION:
Eligible participants for this study must have a diagnosis of probable AD and must have clinically meaningful agitation secondary to AD.

This is a multicenter, randomized, double-dummy, double-blind, placebo-controlled study, consisting of 10 weeks of treatment.

Up to 200 participants will be enrolled at approximately 30-40 centers in the US.

Study medication will be administered orally twice-daily from Day 1 through Day 70. Screening must occur within within approximately 4 weeks prior to randomization. Following screening procedures for assessment of inclusion and exclusion criteria, eligible participants will be randomized into the study.

ELIGIBILITY:
Key Inclusion Criteria:

Diagnosis of probable Alzheimer's disease (AD).

The participant has clinically significant symptoms of agitation secondary to AD, that interfere with daily routine and for which a prescription medication is deemed indicated, in the opinion of the investigator.

Either out-patients or residents of an assisted-living facility or a skilled nursing home.

CGI-S score is ≥ 4 (moderately ill) at screening and baseline.

Mini Mental State Examination (MMSE) score at screening between 8 and 28 (inclusive).

Caregiver who is able and willing to comply with all required study procedures, ensuring that the participant attends all study visits and takes the study medication as instructed. In order to qualify as a caregiver for this study, the individual should spend time with the participant for a minimum of 4 hours on 4 separate days per week.

Key Exclusion Criteria:

Participant has other type of dementia (e.g., vascular dementia, frontotemporal dementia, Parkinson's disease, substance-induced dementia).

Participant with co-existent clinically significant or unstable systemic diseases that could confound the interpretation of the safety results of the study (e.g. malignancy, poorly controlled diabetes, poorly controlled hypertension, unstable pulmonary, renal or hepatic disease, unstable ischemic cardiac disease, dilated cardiomyopathy, certain cardiac conduction abnormalities including QTc prolongation, or unstable valvular heart disease).

Participant with myasthenia gravis.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2012-08-13 (Actual); Primary Completion 2014-07-30 (Actual); Study Completion 2014-07-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (39):
- United States (39):
  - Phoenix, Arizona
  - Sun City, Arizona
  - Fresno, California
  - Fullerton, California
  - Los Angeles, California
  - San Diego, California
  - San Francisco, California
  - Sherman Oaks, California
  - Temecula, California
  - Boynton Beach, Florida
  - Deerfield Beach, Florida
  - Hialeah, Florida
  - Miami, Florida
  - Ocala, Florida
  - Orlando, Florida
  - Sunrise, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Weston, Florida
  - Elk Grove Village, Illinois
  - Las Vegas, Nevada
  - Summit, New Jersey
  - Toms River, New Jersey
  - Orangeburg, New York
  - Rochester, New York
  - White Plains, New York
  - Centerville, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Lakewood, Ohio
  - Allentown, Pennsylvania
  - Reading, Pennsylvania
  - Charleston, South Carolina
  - Houston, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Bennington, Vermont
  - Spokane, Washington

REFERENCES:
- [Background] Cummings JL, Lyketsos CG, Peskind ER, Porsteinsson AP, Mintzer JE, Scharre DW, De La Gandara JE, Agronin M, Davis CS, Nguyen U, Shin P, Tariot PN, Siffert J. Effect of Dextromethorphan-Quinidine on Agitation in Patients With Alzheimer Disease Dementia: A Randomized Clinical Trial. JAMA. 2015 Sep 22-29;314(12):1242-54. doi: 10.1001/jama.2015.10214. PMID 26393847

RESULTS

PARTICIPANT FLOW:
Groups:
- Stage 1: AVP-923: Participants received oral AVP-923 during Stage 1 for 5 consecutive weeks. Participants received AVP-923-20 once daily (QD) in the morning and placebo in the evening (to maintain the blind) during the first week of Stage 1 (Days 1 to 7), AVP-923-20 twice a day (BID) during the next 2 consecutive weeks (Days 8 to 21), and AVP-923-30 BID during the final 2 weeks of Stage 1 (Days 22 to 35).
  (AVP-923-20: 20 milligrams (mg) of dextromethorphan and 10 mg of quinidine; AVP-923-30: 30 mg of dextromethorphan and 10 mg of quinidine)
- Stage 1: Placebo: Participants received matching oral placebo during Stage 1 for 5 consecutive weeks.
- AVP-923 in Stage 1/AVP-923 in Stage 2: Participants received oral AVP-923 during Stage 1 for 5 consecutive weeks. Participants received AVP-923-20 QD in the morning and placebo in the evening (to maintain the blind) during the first week of Stage 1 (Days 1 to 7), AVP-923-20 BID during the next 2 consecutive weeks (Days 8 to 21), and AVP-923-30 BID during the final 2 weeks of Stage 1 (Days 22 to 35). Participants who completed Stage 1 were eligible to participate in Stage 2 of the study. Participants continued to receive AVP-923-30 BID for the entire 5-week duration of Stage 2. Participants received AVP-923-20 QD in the morning and placebo in the evening (to maintain the blind) during the first week of Stage 2 (Days 36 to 42), AVP-923-20 BID during the next 2 consecutive weeks (Days 43 to 56), and AVP-923-30 BID during the final 2 weeks of Stage 2 (Days 57 to 70).
- Placebo in Stage 1/AVP-923 in Stage 2: Participants received matching oral placebo during Stage 1 for 5 consecutive weeks. Participants who completed Stage 1 were eligible to participate in Stage 2 of the study. Participants who were randomized to placebo in Stage 1 were stratified (based on their clinical response during Stage 1) into two subgroups (responders or non-responders) and were re-randomized to receive AVP-923 in Stage 2. Participants received AVP-923-20 QD in the morning and placebo in the evening (to maintain the blind) during the first week of Stage 2 (Days 36 to 42), AVP-923-20 BID during the next 2 consecutive weeks (Days 43 to 56), and AVP-923-30 BID during the final 2 weeks of Stage 2 (Days 57 to 70).
- Placebo in Stage 1/Placebo in Stage 2: Participants received matching oral placebo during Stage 1 for 5 consecutive weeks. Participants who completed Stage 1 were eligible to participate in Stage 2 of the study. Participants who were randomized to placebo in Stage 1 were stratified (based on their clinical response during Stage 1) into two subgroups (responders or non-responders) and were re-randomized to receive matching placebo BID throughout Stage 2.
Period: Stage 1 (5 Weeks)
Arm/Group | Stage 1: AVP-923 | Stage 1: Placebo | AVP-923 in Stage 1/AVP-923 in Stage 2 | Placebo in Stage 1/AVP-923 in Stage 2 | Placebo in Stage 1/Placebo in Stage 2
Started | 93 | 127 | 0 | 0 | 0
Completed | 83 | 119 | 0 | 0 | 0
Not Completed | 10 | 8 | 0 | 0 | 0
Not completed — Advised Not to Take Study Medication | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 5 | 3 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 2 | 3 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Parent/Guardian | 0 | 2 | 0 | 0 | 0
Period: Stage 2 (5 Weeks)
Arm/Group | Stage 1: AVP-923 | Stage 1: Placebo | AVP-923 in Stage 1/AVP-923 in Stage 2 | Placebo in Stage 1/AVP-923 in Stage 2 | Placebo in Stage 1/Placebo in Stage 2
Started | 0 | 0 | 83 | 59 | 60
Completed | 0 | 0 | 80 | 55 | 59
Not Completed | 0 | 0 | 3 | 4 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 2 | 1
Not completed — Unable to Return to Site: Rehabilitation | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline data were collected in members of the Stage 1 modified Intent-to-Treat Population, comprised of all participants randomized in Stage 1 who had at least one post-Baseline Neuropsychiatric Inventory (NPI) agitation/aggression score in Stage 1.
Groups:
- AVP-923: Participants received oral AVP-923 during Stage 1 for 5 consecutive weeks. Participants received AVP-923-20 once daily (QD) in the morning and placebo in the evening (to maintain the blind) during the first week of Stage 1 (Days 1 to 7), AVP-923-20 twice a day (BID) during the next 2 consecutive weeks (Days 8 to 21), and AVP-923-30 BID during the final 2 weeks of Stage 1 (Days 22 to 35).
- Placebo: Participants received matching oral placebo during Stage 1 for 5 consecutive weeks.
- Total: Total of all reporting groups
Arm/Group | AVP-923 | Placebo | Total
Number analyzed (Participants) | 93 | 125 | 218
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.8 (8.01) | 77.6 (7.19) | 77.7 (7.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 74 | 126
  Male | 41 | 51 | 92
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 5 | 6 | 11
  White | 84 | 116 | 200
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in the Neuropsychiatric Inventory (NPI) Agitation/Aggression Domain Score From Day 1 (Stage 1 Baseline) to Day 36 (Stage 2 Baseline) and From Day 36 to Day 70
Description: The NPI is a retrospective interview covering 12 neuropsychiatric symptom domains and is used to evaluate psychopathology, neuropsychiatric manifestations, and caregiver distress. The Agitation/Aggression domain was designed to collect information on the behavioral aspects of agitation/aggression in participants with probable Alzheimer's Disease (AD) and clinically meaningful agitation secondary to AD. Each NPI domain is rated by the caregiver for symptom frequency and severity. Symptom frequency is rated as: 1, occasionally; 2, often; 3, frequently; 4, very frequently. Symptom severity is rated as: 1, mild; 2, moderate; 3, marked. The total domain score is calculated as the frequency score multiplied by the severity score and thus ranges from 1 to 12. A higher score represents worsening symptoms. Change from Baseline is calculated as the post-Baseline score minus the Baseline score. Data are reported for only those participants contributing data to the analysis.
Time Frame: Day 1 (Stage 1 Baseline); Day 36 (Stage 2 Baseline); Day 70
Population: Stage 1 modified Intent-to-Treat (mITT) Population: all participants randomized in Stage 1 who had at least one post-Baseline NPI agitation/aggression score in Stage 1. Stage 2 mITT Population: all placebo non-responders from Stage 1 who were re-randomized in Stage 2 and had at least one post-Week 4 NPI agitation/aggression score in Stage 2
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo: All participants randomized to receive placebo in Stage 1, and all placebo non-responders re-randomized at Stage 2 to placebo
- AVP-923: All participants randomized to receive AVP-923 in Stage 1, and all placebo non-responders re-randomized at Stage 2 to AVP-923.
Arm/Group | Placebo | AVP-923
Number analyzed (Participants) | 125 | 93
score on a scale
  Day 36 | -1.7 (3.10) | -3.3 (2.98)
  Day 70: number analyzed (Participants) | 45 | 44
  Day 70 | -0.8 (3.59) | -2.0 (3.19)
Statistical Analysis 1: Comparison: Placebo vs AVP-923; Test type: Superiority; p <= 0.001, ANCOVA; Sequential Parallel Comparison Design (SPCD): data from the Stages 1 and 2 are analyzed together using the mITT Population; Ordinary Least Squares (OLS) Z-statistic = -1.50
Statistical Analysis 2: Comparison: Placebo vs AVP-923; Test type: Superiority; ANCOVA Least Squares Mean Difference = -1.50 — Day 36
Statistical Analysis 3: Comparison: Placebo vs AVP-923; Test type: Superiority; ANCOVA Least Squares Mean Difference = -1.59 — Day 70

2. Secondary Outcome: Number of Participants With the Indicated Type of Adverse Event
Description: Treatment-emergent adverse events (TEAEs) are defined as AEs that first occurred, or worsened, after the first dose of study medication and within 30 days after the permanent discontinuation of the study medication (first dose date ≤ AE start date ≤ date of last dose + 30 days)
Time Frame: up to Week 10
Population: Safety Population: all randomized participants who received at least one dose of study treatment
Measure: Count of Participants; unit: Participants
Groups:
- All AVP-923: Participants received AVP-923 in either stage.
- Placebo: Participants received placebo in either stage.
Arm/Group | All AVP-923 | Placebo
Number analyzed (Participants) | 152 | 127
Participants
  Participants with ≥ 1 TEAE | 93 | 55
  Participants with discontinuations due to a TEAE | 8 | 4
  Participants who died | 0 | 0

3. Secondary Outcome: Change in the Total NPI Score From Day 1 (Stage 1 Baseline) to Day 36 (Stage 2 Baseline) and From Day 36 to Day 70
Description: The NPI is a retrospective interview covering 12 neuropsychiatric symptom domains and is used to evaluate psychopathology, neuropsychiatric manifestations, and caregiver distress. Each NPI domain is rated by the caregiver for symptom frequency and severity. Symptom frequency is rated as: 1, occasionally; 2, often; 3, frequently; 4, very frequently. Symptom severity is rated as: 1, mild; 2, moderate; 3, marked. The total domain score is calculated as the frequency score multiplied by the severity score and thus ranges from 1 to 12. The total score is calculated as a sum of all 12 domain scores and thus ranges from 12 to 144. A higher score represents worsening symptoms. Change from Baseline is calculated as the post-Baseline score minus the Baseline score.
Time Frame: Day 1 (Stage 1 Baseline); Day 36 (Stage 2 Baseline); Day 70
Population: Stage 1 and Stage 2 mITT Population. Data are reported for only those participants contributing data to the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | AVP-923
Number analyzed (Participants) | 125 | 93
score on a scale
  Day 36 | -8.5 (14.35) | -13.5 (17.48)
  Day 70: number analyzed (Participants) | 45 | 44
  Day 70 | -2.5 (11.82) | -6.0 (2.48)
Statistical Analysis 1: Comparison: Placebo vs AVP-923; Test type: Superiority; p = 0.014, ANCOVA; SPCD: data from the Stages 1 and 2 are analyzed together using the mITT Population; OLS Z-statistic = -2.46
Statistical Analysis 2: Comparison: Placebo vs AVP-923; Test type: Superiority; ANCOVA Least Squares Mean Difference = -4.20; Day 36
Statistical Analysis 3: Comparison: Placebo vs AVP-923; Test type: Superiority; ANCOVA Least Squares Mean Difference = -3.78 — Day 70

4. Secondary Outcome: Change in the Individual NPI Domain Scores From Day 1 (Stage 1 Baseline) to Day 36 (Stage 2 Baseline) and From Day 36 to Day 70
Description: The NPI is a retrospective interview covering 12 neuropsychiatric symptom domains and is used to evaluate psychopathology, neuropsychiatric manifestations, and caregiver distress. Each NPI domain is rated by the caregiver for symptom frequency and severity. Symptom frequency is rated as: 1, occasionally; 2, often; 3, frequently; 4, very frequently. Symptom severity is rated as: 1, mild; 2, moderate; 3, marked. The total domain score is calculated as the frequency score multiplied by the severity score and thus ranges from 1 to 12. A higher score represents worsening symptoms. Change from Baseline is calculated as the post-Baseline score minus the Baseline score. Sleep/nighttime behavior disorders = S/NB disorders.
Time Frame: Day 1 (Stage 1 Baseline); Day 36 (Stage 2 Baseline); Day 70
Population: Stage 1 and Stage 2 mITT Population. Data are reported for only those participants contributing data to the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | AVP-923
Number analyzed (Participants) | 125 | 93
score on a scale
  Day 36, Delusions | -0.6 (2.93) | -0.8 (2.89)
  Day 36, Hallucinations | -0.1 (1.68) | 0.2 (1.76)
  Day 36, Depression/dysphoria | -1.0 (2.89) | -0.9 (2.49)
  Day 36, Anxiety | -1.2 (3.69) | -0.6 (3.21)
  Day 36, Euphoria/elation | -0.1 (1.27) | -0.3 (1.85)
  Day 36, Apathy/indifference | -0.5 (3.69) | -0.9 (4.11)
  Day 36, Disinhibition | -0.7 (3.04) | -0.9 (3.46)
  Day 36, Irritability/lability | -1.2 (3.23) | -2.2 (4.08)
  Day 36, Aberrant motor behavior | -0.4 (3.95) | -1.2 (3.98)
  Day 36, S/NB disorders | -0.1 (2.50) | -1.0 (3.82)
  Day 36, Appetite/eating changes | -1.2 (3.25) | -1.2 (3.68)
  Day 70, Delusions: number analyzed (Participants) | 45 | 44
  Day 70, Delusions | -0.7 (3.09) | 0.1 (3.17)
  Day 70, Hallucinations: number analyzed (Participants) | 45 | 44
  Day 70, Hallucinations | -0.4 (1.60) | -0.1 (2.03)
  Day 70, Depression/dysphoria: number analyzed (Participants) | 45 | 44
  Day 70, Depression/dysphoria | 0.2 (2.36) | 0.2 (2.20)
  Day 70, Anxiety: number analyzed (Participants) | 45 | 44
  Day 70, Anxiety | -0.3 (2.89) | -1.0 (2.76)
  Day 70, Euphoria/elation: number analyzed (Participants) | 45 | 93
  Day 70, Euphoria/elation | -0.0 (1.25) | -0.2 (0.95)
  Day 70, Apathy/indifference: number analyzed (Participants) | 45 | 44
  Day 70, Apathy/indifference | 0.4 (1.96) | -0.5 (3.43)
  Day 70, Disinhibition: number analyzed (Participants) | 45 | 44
  Day 70, Disinhibition | -0.8 (2.51) | -0.8 (2.67)
  Day 70, Irritability/lability: number analyzed (Participants) | 45 | 44
  Day 70, Irritability/lability | -0.7 (3.71) | -1.0 (3.40)
  Day 70, Aberrant motor behavior: number analyzed (Participants) | 45 | 44
  Day 70, Aberrant motor behavior | 0.4 (3.15) | -0.8 (2.52)
  Day 70, S/NB disorders: number analyzed (Participants) | 45 | 44
  Day 70, S/NB disorders | -0.1 (2.04) | 0.0 (2.46)
  Day 70, Appetite/eating changes: number analyzed (Participants) | 45 | 44
  Day 70, Appetite/eating changes | 0.4 (2.28) | 0.1 (2.73)
Statistical Analysis 1: Comparison: Placebo vs AVP-923; Test type: Superiority; p = 0.444, ANCOVA; Delusions Domain. SPCD: data from the Stages 1 and 2 are analyzed together using the mITT Population; OLS Z-statistic = 0.77
Statistical Analysis 2: Comparison: Placebo vs AVP-923; Test type: Superiority; ANCOVA Least Squares Mean Difference = -0.27 — Delusions Domain; Day 36
Statistical Analysis 3: Comparison: Placebo vs AVP-923; Test type: Superiority; ANCOVA Least Squares Mean Difference = 0.78 — Delusions Domain; Day 70
Statistical Analysis 4: Comparison: Placebo vs AVP-923; Test type: Superiority; p = 0.861, ANCOVA; Hallucinations Domain. SPCD: data from the Stages 1 and 2 are analyzed together using the mITT Population; OLS Z-statistic = -0.18
Statistical Analysis 5: Comparison: Placebo vs AVP-923; Test type: Superiority; ANCOVA Least Squares Mean Difference = -0.29 — Hallucinations Domain; Day 36
Statistical Analysis 6: Comparison: Placebo vs AVP-923; Test type: Superiority; ANCOVA Least Squares Mean Difference = 0.22 — Hallucinations Domain; Day 70
Statistical Analysis 7: Comparison: Placebo vs AVP-923; Test type: Superiority; p = 0.749, ANCOVA; Depression/Dysphoria Domain. SPCD: data from the Stages 1 and 2 are analyzed together using the mITT Population; OLS Z-statistic = -0.32
Statistical Analysis 8: Comparison: Placebo vs AVP-923; Test type: Superiority; ANCOVA Least Squares Mean Difference = -0.07 — Depression/Dysphoria Domain; Day 36
Statistical Analysis 9: Comparison: Placebo vs AVP-923; Test type: Superiority; ANCOVA Least Squares Mean Difference = -0.10 — Depression/Dysphoria Domain; Day 70
Statistical Analysis 10: Comparison: Placebo vs AVP-923; Test type: Superiority; p = 0.416, ANCOVA; Anxiety Domain. SPCD: data from the Stages 1 and 2 are analyzed together using the mITT Population; OLS Z-statistic = -0.81
Statistical Analysis 11: Comparison: Placebo vs AVP-923; Test type: Superiority; ANCOVA Least Squares Mean Difference = 0.28 — Anxiety Domain; Day 36
Statistical Analysis 12: Comparison: Placebo vs AVP-923; Test type: Superiority; ANCOVA Least Squares Mean Difference = -0.81 — Anxiety Domain
Statistical Analysis 13: Comparison: Placebo vs AVP-923; Test type: Superiority; p = 0.287, ANCOVA; Euphoria/Elation Domain. SPCD: data from the Stages 1 and 2 are analyzed together using the mITT Population; OLS Z-statistic = -1.07
Statistical Analysis 14: Comparison: Placebo vs AVP-923; Test type: Superiority; ANCOVA Least Squares Mean Difference = 0.04 — Euphoria/Elation Domain; Day 36
Statistical Analysis 15: Comparison: Placebo vs AVP-923; Test type: Superiority; ANCOVA Least Squares Mean Difference = -0.34 — Euphoria/Elation Domain; Day 70
Statistical Analysis 16: Comparison: Placebo vs AVP-923; Test type: Superiority; p = 0.191, ANCOVA; Apathy/Indifference Domain. SPCD: data from the Stages 1 and 2 are analyzed together using the mITT Population; OLS Z-statistic = -1.31
Statistical Analysis 17: Comparison: Placebo vs AVP-923; Test type: Superiority; ANCOVA Least Squares Mean Difference = -0.16 — Apathy/Indifference Domain; Day 36
Statistical Analysis 18: Comparison: Placebo vs AVP-923; Test type: Superiority; ANCOVA Least Squares Mean Difference = -0.77 — Apathy/Indifference Domain; Day 36
Statistical Analysis 19: Comparison: Placebo vs AVP-923; Test type: Superiority; p = 0.271, ANCOVA; Disinhibition Domain. SPCD: data from the Stages 1 and 2 are analyzed together using the mITT Population; OLS Z-statistic = -1.10
Statistical Analysis 20: Comparison: Placebo vs AVP-923; Test type: Superiority; ANCOVA Least Squares Mean Difference = -0.22 — Disinhibition Domain; Day 36
Statistical Analysis 21: Comparison: Placebo vs AVP-923; Test type: Superiority; ANCOVA Least Squares Mean Difference = -0.37 — Disinhibition Domain; Day 70
Statistical Analysis 22: Comparison: Placebo vs AVP-923; Test type: Superiority; p = 0.029, ANCOVA; Irritability/Lability Domain. SPCD: data from the Stages 1 and 2 are analyzed together using the mITT Population; OLS Z-statistic = -2.18
Statistical Analysis 23: Comparison: Placebo vs AVP-923; Test type: Superiority; ANCOVA Least Squares Mean Difference = -0.70 — Irritability/Lability Domain; Day 36
Statistical Analysis 24: Comparison: Placebo vs AVP-923; Test type: Superiority; ANCOVA Least Squares Mean Difference = -0.93 — Irritability/Lability Domain; Day 70
Statistical Analysis 25: Comparison: Placebo vs AVP-923; Test type: Superiority; p = 0.027, ANCOVA; Aberrant Motor Behavior Domain. SPCD: data from the Stages 1 and 2 are analyzed together using the mITT Population; OLS Z-statistic = -2.21
Statistical Analysis 26: Comparison: Placebo vs AVP-923; Test type: Superiority; ANCOVA Least Squares Mean Difference = -0.38 — Aberrant Motor Behavior Domain; Day 36
Statistical Analysis 27: Comparison: Placebo vs AVP-923; Test type: Superiority; ANCOVA Least Squares Mean Difference = -1.22 — Aberrant Motor Behavior Domain; Day 70
Statistical Analysis 28: Comparison: Placebo vs AVP-923; Test type: Superiority; p = 0.274, ANCOVA; Sleep/Nighttime Behavior Disorders Domain. SPCD: data from the Stages 1 and 2 are analyzed together using the mITT Population; OLS Z-statistic = -1.09
Statistical Analysis 29: Comparison: Placebo vs AVP-923; Test type: Superiority; ANCOVA Least Squares Mean Difference = -0.57 — Sleep/Nighttime Behavior disorders Domain; Day 36
Statistical Analysis 30: Comparison: Placebo vs AVP-923; Test type: Superiority; ANCOVA Least Squares Mean Difference = -0.08 — Sleep/Nighttime Behavior disorders Domain; Day 70
Statistical Analysis 31: Comparison: Placebo vs AVP-923; Test type: Superiority; p = 0.513, ANCOVA; Appetite/Eating Changes Domain. SPCD: data from the Stages 1 and 2 are analyzed together using the mITT Population; OLS Z-statistic = -0.65
Statistical Analysis 32: Comparison: Placebo vs AVP-923; Test type: Superiority; ANCOVA Least Squares Mean Difference = -0.16 — Appetite/Eating Changes Domain; Day 36
Statistical Analysis 33: Comparison: Placebo vs AVP-923; Test type: Superiority; ANCOVA Least Squares Mean Difference = -0.24 — Appetite/Eating Changes Domain; Day 70

5. Secondary Outcome: Change in the Sum of the Agitation/Aggression, Irritability/Lability, Disinhibition, and Aberrant Motor Behavior NPI Domain (NPI4D) Score From Day 1 (Stage 1 Baseline) to Day 36 (Stage 2 Baseline) and From Day 36 to Day 70
Description: The NPI is a retrospective interview covering 12 neuropsychiatric symptom domains and is used to evaluate psychopathology, neuropsychiatric manifestations, and caregiver distress. Each NPI domain is rated by the caregiver for symptom frequency and severity. Symptom frequency is rated as: 1, occasionally; 2, often; 3, frequently; 4, very frequently. Symptom severity is rated as: 1, mild; 2, moderate; 3, marked. The total domain score is calculated as the frequency score multiplied by the severity score and thus ranges from 1 to 12. The NPI4D score is the sum of the Agitation/Aggression, Irritability/Lability, Disinhibition, and Aberrant Motor Behavior domain scores, and thus ranges from 4 to 48. A higher score represents worsening symptoms. Change from Baseline is calculated as the post-Baseline score minus the Baseline score.
Time Frame: Day 1 (Stage 1 Baseline); Day 36 (Stage 2 Baseline); Day 70
Population: Stage 1 and Stage 2 mITT Populations. Data are reported for only those participants contributing data to the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | AVP-923
Number analyzed (Participants) | 125 | 93
score on a scale
  Day 36 | -4.0 (8.24) | -7.6 (9.08)
  Day 70: number analyzed (Participants) | 45 | 44
  Day 70 | -1.9 (7.65) | -4.6 (7.31)
Statistical Analysis 1: Comparison: Placebo vs AVP-923; Test type: Superiority; p <= 0.001, ANCOVA; SPCD: data from the Stages 1 and 2 are analyzed together using the mITT Population; OLS Z-statistic = -3.53
Statistical Analysis 2: Comparison: Placebo vs AVP-923; Test type: Superiority; ANCOVA Least Squares Mean Difference = -3.01 — Day 36
Statistical Analysis 3: Comparison: Placebo vs AVP-923; Test type: Superiority; ANCOVA Least Squares Mean Difference = -3.49 — Day 70

6. Secondary Outcome: Change in the Sum of the Agitation/Aggression, Irritability/Lability, Anxiety, and Aberrant Motor Behavior NPI Domain (NPI4A) Score From Day 1 (Stage 1 Baseline) to Day 36 (Stage 2 Baseline) and From Day 36 to Day 70
Description: The NPI is a retrospective interview covering 12 neuropsychiatric symptom domains and is used to evaluate psychopathology, neuropsychiatric manifestations, and caregiver distress. Each NPI domain is rated by the caregiver for symptom frequency and severity. Symptom frequency is rated as: 1, occasionally; 2, often; 3, frequently; 4, very frequently. Symptom severity is rated as: 1, mild; 2, moderate; 3, marked. The total domain score is calculated as the frequency score multiplied by the severity score and thus ranges from 1 to 12. The NPI4A score is the sum of the Agitation/Aggression, Irritability/Lability, Anxiety, and Aberrant Motor Behavior domain scores, and thus ranges from 4 to 48. A higher score represents worsening symptoms. Change from Baseline is calculated as the post-Baseline score minus the Baseline score.
Time Frame: Day 1 (Stage 1 Baseline); Day 36 (Stage 2 Baseline); Day 70
Population: Stage 1 and Stage 2 mITT Populations. Data are reported for only those participants contributing data to the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | AVP-923
Number analyzed (Participants) | 125 | 93
score on a scale
  Day 36 | -4.5 (8.53) | -7.3 (9.08)
  Day 70: number analyzed (Participants) | 45 | 44
  Day 70 | -1.4 (7.94) | -4.8 (7.05)
Statistical Analysis 1: Comparison: Placebo vs AVP-923; Test type: Superiority; p = 0.001, ANCOVA; SPCD: data from the Stages 1 and 2 are analyzed together using the mITT Population; OLS Z-statistic = -3.34
Statistical Analysis 2: Comparison: Placebo vs AVP-923; Test type: Superiority; ANCOVA Least Squares Mean Difference = -2.41 — Day 36
Statistical Analysis 3: Comparison: Placebo vs AVP-923; Test type: Superiority; ANCOVA Least Squares Mean Difference = -3.94 — Day 70

7. Secondary Outcome: Change in the Total Neuropsychiatric Inventory-Caregiver Distress Score (NPI-CDS) From Day 1 (Stage 1 Baseline) to Day 36 (Stage 2 Baseline) and From Day 36 to Day 70
Description: The NPI is a retrospective interview covering 12 neuropsychiatric symptom domains and is used to evaluate psychopathology, neuropsychiatric manifestations, and caregiver distress. For each domain, the caregiver is asked to rate how emotionally distressing they find the symptom behavior on the following scale: 0, not at all; 1, minimally; 2, mildly; 3, moderately; 4, severely; 5, very severely or extremely. The total NPI-CDS score is calculated as the sum of all 12 domain scores and thus ranges from 0 to 60. A higher score represents increased distress. Change from Baseline is calculated as the post-Baseline score minus the Baseline score.
Time Frame: Day 1 (Stage 1 Baseline); Day 36 (Stage 2 Baseline); Day 70
Population: Stage 1 and Stage 2 mITT Populations. Data are reported for only those participants contributing data to the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | AVP-923
Number analyzed (Participants) | 125 | 93
score on a scale
  Day 36 | -3.6 (6.64) | -6.6 (7.81)
  Day 70: number analyzed (Participants) | 45 | 44
  Day 70 | -2.0 (5.74) | -2.6 (5.52)
Statistical Analysis 1: Comparison: Placebo vs AVP-923; Test type: Superiority; p = 0.014, ANCOVA; SPCD: data from the Stages 1 and 2 are analyzed together using the mITT Population; OLS Z-statistic = -2.46
Statistical Analysis 2: Comparison: Placebo vs AVP-923; Test type: Superiority; ANCOVA Least Squares Mean Difference = -2.65 — Day 36
Statistical Analysis 3: Comparison: Placebo vs AVP-923; Test type: Superiority; ANCOVA Least Squares Mean Difference = -1.01; Day 70

8. Secondary Outcome: Change in the NPI-CDS for the Agitation/Aggression Domain From Day 1 (Stage 1 Baseline) to Day 36 (Stage 2 Baseline) and From Day 36 to Day 70
Description: The NPI is a retrospective interview covering 12 neuropsychiatric symptom domains and is used to evaluate psychopathology, neuropsychiatric manifestations, and caregiver distress. For the Agitation/Aggression domain, the caregiver is asked to rate how emotionally distressing they find the symptom behavior on the following scale: 0, not at all; 1, minimally; 2, mildly; 3, moderately; 4, severely; 5, very severely or extremely. A higher score represents increased distress. Change from Baseline is calculated as the post-Baseline score minus the Baseline score.
Time Frame: Day 1 (Stage 1 Baseline); Day 36 (Stage 2 Baseline); Day 70
Population: Stage 1 and Stage 2 mITT Populations. Data are reported for only those participants contributing data to the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | AVP-923
Number analyzed (Participants) | 125 | 93
score on a scale
  Day 36 | -0.6 (1.32) | -1.4 (1.54)
  Day 70: number analyzed (Participants) | 45 | 44
  Day 70 | -0.7 (1.38) | -0.5 (1.44)
Statistical Analysis 1: Comparison: Placebo vs AVP-923; Test type: Superiority; p = 0.010, ANCOVA; SPCD: data from the Stages 1 and 2 are analyzed together using the mITT Population; OLS Z-statistic = -2.57
Statistical Analysis 2: Comparison: Placebo vs AVP-923; Test type: Superiority; ANCOVA Least Squares Mean Difference = -0.68 — Day 36
Statistical Analysis 3: Comparison: Placebo vs AVP-923; Test type: Superiority; ANCOVA Least Squares Mean Difference = -0.20 — Day 70

9. Secondary Outcome: Change in the NPI-CDS NPI4D Score From Day 1 (Stage 1 Baseline) to Day 36 (Stage 2 Baseline) and From Day 36 to Day 70
Description: The NPI is a retrospective interview covering 12 neuropsychiatric symptom domains and is used to evaluate psychopathology, neuropsychiatric manifestations, and caregiver distress. For the NPI4D NPI-CDS score, the caregiver is asked to rate how emotionally distressing they find the symptom behavior (for the Agitation/Aggression, Irritability/Lability, Disinhibition, and Aberrant Motor Behavior domains) on the following scale: 0, not at all; 1, minimally; 2, mildly; 3, moderately; 4, severely; 5, very severely or extremely. The NPI4D NPI-CDS score ranges from 0 to 20. A higher score represents increased distress. Change from Baseline is calculated as the post-Baseline score minus the Baseline score.
Time Frame: Day 1 (Stage 1 Baseline); Day 36 (Stage 2 Baseline); Day 70
Population: Stage 1 and Stage 2 mITT Populations. Data are reported for only those participants contributing data to the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | AVP-923
Number analyzed (Participants) | 125 | 93
score on a scale
  Day 36 | -1.5 (3.39) | -3.3 (4.11)
  Day 70: number analyzed (Participants) | 45 | 44
  Day 70 | -1.2 (3.08) | -1.8 (3.12)
Statistical Analysis 1: Comparison: Placebo vs AVP-923; Test type: Superiority; p = 0.002, ANCOVA; SPCD: data from the Stages 1 and 2 are analyzed together using the mITT Population; OLS Z-statistic = -3.08
Statistical Analysis 2: Comparison: Placebo vs AVP-923; Test type: Superiority; ANCOVA Least Squares Mean Difference = -1.56 — Day 36
Statistical Analysis 3: Comparison: Placebo vs AVP-923; Test type: Superiority; ANCOVA Least Squares Mean Difference = -0.90 — Day 70

10. Secondary Outcome: Change in the NPI-CDS NPI4A Score From Day 1 (Stage 1 Baseline) to Day 36 (Stage 2 Baseline) and From Day 36 to Day 70
Description: The NPI is a retrospective interview covering 12 neuropsychiatric symptom domains and is used to evaluate psychopathology, neuropsychiatric manifestations, and caregiver distress. For the NPI4A NPI-CDS score, the caregiver is asked to rate how emotionally distressing they find the symptom behavior (for the Agitation/Aggression, Irritability/Lability, Anxiety, and Aberrant Motor Behavior domains) on the following scale: 0, not at all; 1, minimally; 2, mildly; 3, moderately; 4, severely; 5, very severely or extremely. The NPI4A NPI-CDS score ranges from 0 to 20. Change from Baseline is calculated as the post-Baseline score minus the Baseline score.
Time Frame: Day 1 (Stage 1 Baseline); Day 36 (Stage 2 Baseline); Day 70
Population: Stage 1 and Stage 2 mITT Populations. Data are reported for only those participants contributing data to the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | AVP-923
Number analyzed (Participants) | 125 | 93
score on a scale
  Day 36 | -1.7 (3.34) | -3.3 (3.84)
  Day 70: number analyzed (Participants) | 45 | 44
  Day 70 | -1.0 (3.51) | -1.5 (2.70)
Statistical Analysis 1: Comparison: Placebo vs AVP-923; Test type: Superiority; p = 0.008, ANCOVA; SPCD: data from the Stages 1 and 2 are analyzed together using the mITT Population; OLS Z-statistic = -2.66
Statistical Analysis 2: Comparison: Placebo vs AVP-923; Test type: Superiority; ANCOVA Least Squares Mean Difference = -1.43 — Day 36
Statistical Analysis 3: Comparison: Placebo vs AVP-923; Test type: Superiority; ANCOVA Least Squares Mean Difference = -0.75 — Day 70

11. Secondary Outcome: Change in the Caregiver Strain Index (CSI) Score From Day 1 (Stage 1 Baseline) to Day 36 (Stage 2 Baseline) and From Day 36 to Day 70
Description: The CSI is a 13-question tool that is used to measure strain related to care provision and to identify families with potential caregiving concerns. There is at least one item for each of the following major domains: Employment, Financial, Physical, Social, and Time. A 0 (No) to 1 (Yes) scale is used for each of the 13 questions; thus the total score ranges from 0 to 13. Higher scores signify higher stress levels. Positive responses to 7 or more items on the index indicate a greater level of strain. Change from Baseline is calculated as the post-Baseline score minus the Baseline score.
Time Frame: Day 1 (Stage 1 Baseline); Day 36 (Stage 2 Baseline); Day 70
Population: Stage 1 and Stage 2 mITT Populations. Data are reported for only those participants contributing data to the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | AVP-923
Number analyzed (Participants) | 125 | 93
score on a scale
  Day 36 | -0.6 (2.06) | -1.2 (2.37)
  Day 70: number analyzed (Participants) | 45 | 44
  Day 70 | 0.1 (1.88) | -0.2 (1.62)
Statistical Analysis 1: Comparison: Placebo vs AVP-923; Test type: Superiority; p = 0.050, ANCOVA; SPCD: data from the Stages 1 and 2 are analyzed together using the mITT Population; OLS Z-statistic = -1.96
Statistical Analysis 2: Comparison: Placebo vs AVP-923; Test type: Superiority; ANCOVA Least Squares Mean Difference = -0.62 — Day 36
Statistical Analysis 3: Comparison: Placebo vs AVP-923; Test type: Superiority; ANCOVA Least Squares Mean Difference = -0.30 — Day 70

12. Secondary Outcome: Change in the Cornell Scale for Depression in Dementia (CSDD) Score From Day 1 (Stage 1 Baseline) to Day 36 (Stage 2 Baseline) and From Day 36 to Day 70
Description: The CSDD is a 19-item interview specifically developed to assess the signs and symptoms of major depression in participants with dementia. Each of the 19 items is rated for severity on a scale of 0 to 2 (0, absent; 1, mild or intermittent; 2, severe). The total score is calculated as the sum of the item scores and thus ranges from 0 to 38. Higher scores signify more severe depression. Scores above 10 indicate probable major depression. Scores above 18 indicate definite major depression. Scores below 6, as a rule, are associated with the absence of significant depressive symptoms. Change from Baseline is calculated as the post-Baseline score minus the Baseline score.
Time Frame: Day 1 (Stage 1 Baseline); Day 36 (Stage 2 Baseline); Day 70
Population: Stage 1 and Stage 2 mITT Populations. Data are reported for only those participants contributing data to the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | AVP-923
Number analyzed (Participants) | 125 | 93
score on a scale
  Day 36 | 0.6 (3.84) | -1.0 (3.43)
  Day 70: number analyzed (Participants) | 45 | 44
  Day 70 | -0.7 (2.58) | -0.9 (2.93)
Statistical Analysis 1: Comparison: Placebo vs AVP-923; Test type: Superiority; p = 0.020, ANCOVA; SPCD: data from the Stages 1 and 2 are analyzed together using the mITT Population; OLS Z-statistic = -2.33
Statistical Analysis 2: Comparison: Placebo vs AVP-923; Test type: Superiority; ANCOVA Least Squares Mean Difference = -1.57 — Day 36
Statistical Analysis 3: Comparison: Placebo vs AVP-923; Test type: Superiority; ANCOVA Least Squares Mean Difference = -0.18 — Day 70

13. Secondary Outcome: Change in the Mini-Mental State Examination (MMSE) Score From Day 1 (Stage 1 Baseline) to Day 36 (Stage 2 Baseline), as Analyzed by the Specified SPCD Methodology
Description: The MMSE is a brief test that is used to screen for cognitive impairment. The MMSE scale comprises 11 questions or simple tasks concerning orientation, memory, attention, and language to evaluate the participant's cognitive state. The anchor values are not consistent for each task. The MMSE total score is calculated by summing the item scores across all 11 tasks. A participant's total possible MMSE score ranges from 0 to 30 points. Higher scores indicate milder cognitive impairment. Change from Baseline is calculated as the post-Baseline score minus the Baseline score.
Time Frame: Day 1 (Stage 1 Baseline); Day 36 (Stage 2 Baseline); Day 70
Population: Stage 1 and Stage 2 mITT Populations. Data are reported for only those participants contributing data to the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | AVP-923
Number analyzed (Participants) | 125 | 93
score on a scale
  Day 36 | -0.3 (2.77) | 0.2 (3.02)
  Day 70: number analyzed (Participants) | 45 | 44
  Day 70 | -0.5 (2.53) | 0.3 (2.76)
Statistical Analysis 1: Comparison: Placebo vs AVP-923; Test type: Superiority; p = 0.053, ANCOVA; SPCD: data from the Stages 1 and 2 are analyzed together using the mITT Population; OLS Z-statistic = 1.94
Statistical Analysis 2: Comparison: Placebo vs AVP-923; Test type: Superiority; ANCOVA Least Squares Mean Difference = 0.52 — Day 36
Statistical Analysis 3: Comparison: Placebo vs AVP-923; Test type: Superiority; ANCOVA Least Squares Mean Difference = 0.84 — Day 70

14. Secondary Outcome: Change in the Quality of Life-Alzheimer's Disease (QoL-AD) Score From Day 1 (Stage 1 Baseline) to Day 36 (Stage 2 Baseline) and From Day 36 to Day 70
Description: The QoL-AD is a brief, 13-item measure designed specifically to obtain a rating of the participant's quality of life (QoL) from both the participant and the caregiver. It uses simple and straightforward language and responses and includes assessments of the individual's relationships with friends and family, concerns about finances, physical condition, mood, and an overall assessment of life quality. Caregivers complete the measure as a questionnaire about the participants' QoL, whereas participants complete it in interview format about their own QoL. Each of the 13 items is rated on a 4-point scale, with 1 indicating a poor QoL and 4 indicating an excellent QoL. Total scores range from 13 to 52, with a higher score indicating a better QoL. Change from Baseline is calculated as the post-Baseline score minus the Baseline score.
Time Frame: Day 1 (Stage 1 Baseline); Day 36 (Stage 2 Baseline); Day 70
Population: Stage 1 and Stage 2 mITT Populations. Data are reported for only those participants contributing data to the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | AVP-923
Number analyzed (Participants) | 125 | 93
score on a scale
  Day 36, Cargiver | 0.3 (4.66) | 0.4 (4.28)
  Day 70, Caregiver: number analyzed (Participants) | 45 | 44
  Day 70, Caregiver | 0.9 (4.27) | -0.3 (3.93)
  Day 36, Participant | -0.0 (5.18) | 1.3 (6.12)
  Day 70, Participant: number analyzed (Participants) | 45 | 44
  Day 70, Participant | 0.7 (4.26) | 1.5 (5.06)
Statistical Analysis 1: Comparison: Placebo vs AVP-923; Test type: Superiority; p = 0.469, ANCOVA; SPCD: data from the Stages 1 and 2 are analyzed together using the mITT Population; OLS Z-statistic = -0.72 — Caregiver
Statistical Analysis 2: Comparison: Placebo vs AVP-923; Test type: Superiority; ANCOVA Least Squares Mean Difference = 0.28 — Caregiver: Day 36
Statistical Analysis 3: Comparison: Placebo vs AVP-923; Test type: Superiority; ANCOVA Least Squares Mean Difference = -1.06 — Caregiver: Day 70
Statistical Analysis 4: Comparison: Placebo vs AVP-923; Test type: Superiority; p = 0.159, ANCOVA; SPCD: data from the Stages 1 and 2 are analyzed together using the mITT Population; OLS Z-statistic = 1.41 — Participant
Statistical Analysis 5: Comparison: Placebo vs AVP-923; Test type: Superiority; ANCOVA Least Squares Mean Difference = 1.09 — Participant: Day 36
Statistical Analysis 6: Comparison: Placebo vs AVP-923; Test type: Superiority; ANCOVA Least Squares Mean Difference = 0.70 — Participant: Day 70

15. Secondary Outcome: Change in the Alzheimer's Disease Cooperative Study-Activities of Daily Living Inventory (ADCS-ADL) Score From Day 1 (Stage 1 Baseline) to Day 36 (Stage 2 Baseline) and From Day 36 to Day 70
Description: The ADCS-ADL inventory measures basic activities of daily living such as dressing, conversation, eating, bathing, and grooming. The 19-item version, covering mainly basic ADL, is used to assess participants with more severe disabilities. The ADCS-ADL uses a scale from 0 to 54. Lower scores indicate declining ability. Change from Baseline is calculated as the post-Baseline value minus the Baseline value.
Time Frame: Day 1 (Stage 1 Baseline); Day 36 (Stage 2 Baseline); Day 70
Population: Stage 1 and Stage 2 mITT Populations. Data are reported for only those participants contributing data to the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | AVP-923
Number analyzed (Participants) | 125 | 93
score on a scale
  Day 36 | -0.8 (3.89) | -0.9 (4.27)
  Day 70: number analyzed (Participants) | 45 | 44
  Day 70 | -0.6 (3.45) | -2.0 (4.64)
Statistical Analysis 1: Comparison: Placebo vs AVP-923; Test type: Superiority; p = 0.163, ANCOVA; SPCD: data from the Stages 1 and 2 are analyzed together using the mITT Population; OLS Z-statistic = -1.40
Statistical Analysis 2: Comparison: Placebo vs AVP-923; Test type: Superiority; ANCOVA Least Squares Mean Difference = -0.07 — Day 36
Statistical Analysis 3: Comparison: Placebo vs AVP-923; Test type: Superiority; ANCOVA Least Squares Mean Difference = -1.39 — Day 70

16. Secondary Outcome: Change in the NPI Agitation/Aggression Domain Score From Day 1 (Stage 1 Baseline) to Day 8 and Day 22 and From Day 36 (Stage 2 Baseline) to Day 43 and Day 57
Description: The NPI is a retrospective interview covering 12 neuropsychiatric symptom domains and is used to evaluate psychopathology, neuropsychiatric manifestations, and caregiver distress. The Agitation/Aggression domain was designed to collect information on the behavioral aspects of agitation/aggression in participants with probable AD and clinically meaningful agitation secondary to AD. Each NPI domain is rated by the caregiver for symptom frequency and severity. Symptom frequency is rated as: 1, occasionally; 2, often; 3, frequently; 4, very frequently. Symptom severity is rated as: 1, mild; 2, moderate; 3, marked. The total domain score is calculated as the frequency score multiplied by the severity score and thus ranges from 1 to 12. A higher score represents worsening symptoms. Change from Baseline is calculated as the post-Baseline score minus the Baseline score.
Time Frame: Day 1 (Stage 1 Baseline); Days 8 and 22; Day 36 (Stage 2 Baseline); Days 43 and 57
Population: Stage 1 and Stage 2 mITT Populations. Data are reported for only those participants contributing data to the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | AVP-923
Number analyzed (Participants) | 124 | 93
score on a scale
  Day 8 | -1.4 (2.73) | -2.2 (2.93)
  Day 22: number analyzed (Participants) | 121 | 90
  Day 22 | -1.6 (2.86) | -2.7 (3.18)
  Day 43: number analyzed (Participants) | 45 | 44
  Day 43 | -1.3 (2.92) | -0.5 (2.31)
  Day 57: number analyzed (Participants) | 45 | 44
  Day 57 | -1.3 (2.86) | -1.2 (3.12)
Statistical Analysis 1: Comparison: Placebo vs AVP-923; Test type: Superiority; p = 0.279, ANCOVA; SPCD: data from the Stages 1 and 2 are analyzed together using the mITT Population; OLS Z-statistic = -1.08
Statistical Analysis 2: Comparison: Placebo vs AVP-923; Test type: Superiority; ANCOVA Least Squares Mean Difference = -0.76 — Day 8
Statistical Analysis 3: Comparison: Placebo vs AVP-923; Test type: Superiority; ANCOVA Least Squares Mean Difference = -1.02 — Day 22
Statistical Analysis 4: Comparison: Placebo vs AVP-923; Test type: Superiority; ANCOVA Least Squares Mean Difference = 0.74 — Day 43
Statistical Analysis 5: Comparison: Placebo vs AVP-923; Test type: Superiority; ANCOVA Least Squares Mean Difference = -0.05 — Day 57

17. Secondary Outcome: Number of Participants With the Indicated Response on the Alzheimer's Disease Cooperative Study-Clinical Global Impression of Change Rating (mADCS-CGIC) Scale Agitation Domain at Day 36 and Day 70 Compared to Their Response at Day 1 (Stage 1 Baseline)
Description: The intent of the ADCS version of the CGIC is to provide a means to reliably assess the global impression of change from Baseline in a clinical trial. The mADCS-CGIC is a modification of the ADCS-CGIC instrument that focuses specifically on agitation. The participant is asked to rate their impression of change from Baseline as: 1, marked improvement; 2, moderate improvement; 3, minimal improvement; 4, no change; 5, minimal worsening; 6, moderate worsening; 7, marked worsening. Baseline is defined as the last non-missing assessment prior to Stage 1 randomization.
Time Frame: Day 1 (Stage 1 Baseline); Day 36 (Stage 2 Baseline); Day 70
Population: Stage 1 and Stage 2 mITT Populations. Data are reported for only those participants contributing data to the analysis.
Measure: Number; unit: participants
Arm/Group | Placebo | AVP-923
Number analyzed (Participants) | 123 | 88
participants
  Day 36, Marked improvement | 1 | 8
  Day 36, Moderate improvement | 13 | 22
  Day 36, Minimal improvement | 43 | 28
  Day 36, No change | 48 | 22
  Day 36, Minimal worsening | 12 | 7
  Day 36, Moderate worsening | 6 | 1
  Day 36, Marked worsening | 0 | 0
  Day 70, Marked improvement: number analyzed (Participants) | 44 | 42
  Day 70, Marked improvement | 4 | 4
  Day 70, Moderate improvement: number analyzed (Participants) | 44 | 42
  Day 70, Moderate improvement | 5 | 10
  Day 70, Minimal improvement: number analyzed (Participants) | 44 | 42
  Day 70, Minimal improvement | 11 | 10
  Day 70, No change: number analyzed (Participants) | 44 | 42
  Day 70, No change | 14 | 12
  Day 70, Marked worsening: number analyzed (Participants) | 44 | 42
  Day 70, Marked worsening | 9 | 3
  Day 70, Moderate worsening: number analyzed (Participants) | 44 | 42
  Day 70, Moderate worsening | 0 | 3
  Day 70, Minimal worsening: number analyzed (Participants) | 44 | 42
  Day 70, Minimal worsening | 1 | 0
Statistical Analysis 1: Comparison: Placebo vs AVP-923; Test type: Superiority; p = 0.0001, ANCOVA; Odds Ratio (OR) = 2.70, 95% CI 2-sided [1.62 to 4.50] — Day 36
Statistical Analysis 2: Comparison: Placebo vs AVP-923; Test type: Superiority; p = 0.2184, ANCOVA; Odds Ratio (OR) = 1.61, 95% CI 2-sided [0.75 to 3.43] — Day 70

18. Secondary Outcome: Number of Participants With the Indicated Response on the mADCS-CGIC Scale Agitation Domain at Day 70 Compared to Their Response at Day 36 (Stage 2 Baseline)
Description: The intent of the ADCS version of the CGIC is to provide a means to reliably assess the global impression of change from Baseline in a clinical trial. The mADCS-CGIC is a modification of the ADCS-CGIC instrument that focuses specifically on agitation. The participant is asked to rate their impression of change from Baseline as: 1, marked improvement; 2, moderate improvement; 3, minimal improvement; 4, no change; 5, minimal worsening; 6, moderate worsening; 7, marked worsening. For placebo non-responders re-randomized to AVP-923 or placebo at Stage 2, Baseline is defined as the last non-missing assessment prior to Stage 2 re-randomization.
Time Frame: Day 36 (Stage 2 Baseline); Day 70
Population: Stage 2 mITT Population. Data are reported for only those participants contributing data to the analysis.
Measure: Number; unit: participants
Arm/Group | Placebo | AVP-923
Number analyzed (Participants) | 42 | 42
participants
  Marked improvement | 4 | 0
  Moderate improvement | 2 | 11
  Minimal improvement | 8 | 15
  No change | 19 | 11
  Marked worsening | 6 | 4
  Moderate worsening | 2 | 1
  Minimal worsening | 1 | 0
Statistical Analysis 1: Comparison: Placebo vs AVP-923; Test type: Superiority; p = 0.0266, ANCOVA; Odds Ratio (OR) = 2.45, 95% CI 2-sided [1.11 to 5.42]

19. Secondary Outcome: Number of Participants With the Indicated Categorical Response on the Patient Global Impression of Change (PGI-C) for the Caregiver Domain at Day 36 (Stage 2 Baseline) and Day 70 Compared to Their Response at Day 1 (Stage 1 Baseline)
Description: The PGI-C uses a 7-point scale to assess treatment response and to rate the global impression of clinical change in a participant's agitation. The participant is asked to rate their impression of change from Baseline as: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; 7, very much worse. Baseline is defined as the last non-missing assessment prior to Stage 1 randomization.
Time Frame: Day 1 (Stage 1 Baseline); Day 36 (Stage 2 Baseline); Day 70
Population: Stage 1 and Stage 2 mITT Populations. Data are reported for only those participants contributing data to the analysis.
Measure: Number; unit: participants
Arm/Group | Placebo | AVP-923
Number analyzed (Participants) | 123 | 88
participants
  Day 36, Very much improved | 2 | 10
  Day 36, Much improved | 23 | 24
  Day 36, Minimally improved | 30 | 20
  Day 36, No change | 40 | 20
  Day 36, Minimally worse | 23 | 13
  Day 36, Much worse | 4 | 1
  Day 36, Very much worse | 1 | 0
  Day 70, Very much improved: number analyzed (Participants) | 44 | 43
  Day 70, Very much improved | 3 | 3
  Day 70, Much improved: number analyzed (Participants) | 44 | 43
  Day 70, Much improved | 4 | 10
  Day 70, Minimally improved: number analyzed (Participants) | 44 | 43
  Day 70, Minimally improved | 11 | 14
  Day 70, No change: number analyzed (Participants) | 44 | 43
  Day 70, No change | 13 | 10
  Day 70, Minimally worse: number analyzed (Participants) | 44 | 43
  Day 70, Minimally worse | 9 | 4
  Day 70, Much worse: number analyzed (Participants) | 44 | 43
  Day 70, Much worse | 4 | 2
  Day 70, Very much worse: number analyzed (Participants) | 44 | 43
  Day 70, Very much worse | 0 | 0
Statistical Analysis 1: Comparison: Placebo vs AVP-923; Test type: Superiority; p = 0.002, ANCOVA; Odds Ratio (OR) = 2.16, 95% CI 2-sided [1.31 to 3.55] — Day 36
Statistical Analysis 2: Comparison: Placebo vs AVP-923; Test type: Superiority; p = 0.031, ANCOVA; Odds Ratio (OR) = 2.32, 95% CI 2-sided [1.08 to 5.00] — Day 70

20. Secondary Outcome: Number of Participants With the Indicated Categorical Response on the PGI-C for the Caregiver Domain at Day 70 Compared to Their Response at Day 1 (Stage 1 Baseline)
Description: The PGI-C uses a 7-point scale to assess treatment response and to rate the global impression of clinical change in a participant's agitation. The participant is asked to rate their impression of change from Baseline as: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; 7, very much worse. For placebo non-responders re-randomized to AVP-923 or placebo at Stage 2, Baseline is defined as the last non-missing assessment prior to Stage 2 re-randomization.
Time Frame: Day 1 (Stage 1 Baseline); Day 70
Population: Only AVP-923/only placebo ITT Subset
Measure: Number; unit: participants
Arm/Group | Placebo | AVP-923
Number analyzed (Participants) | 59 | 81
participants
  Very much improved | 5 | 9
  Much improved | 9 | 26
  Minimally improved | 17 | 25
  No change | 14 | 13
  Minimally worse | 10 | 5
  Much worse | 4 | 3
  Very much worse | 0 | 0
Statistical Analysis 1: Comparison: Placebo vs AVP-923; Test type: Superiority; p = 0.0048, ANCOVA; Odds Ratio (OR) = 2.41, 95% CI 2-sided [1.31 to 4.46]

21. Secondary Outcome: Number of Participants With the Indicated Change in the Concomitant Use of Allowed Psychotropic Drugs Compared to Their Baseline Use
Description: Concomitant medications (CMs) are defined as non-study medications with a start date on or before the final study visit, and that were either ongoing at the end of the study or had a stop date on or after the date of first dose of study drug. Drugs for the treatment of AD (e.g., donepezil, rivastigmine, galantamine, memantine) were allowed when administered at stable dose for at least 2 months prior to randomization. Concomitant use of the following medications was allowed, provided the participant had been on a stable dose for at least 1 month prior to randomization and remained stable throughout the study: medications for agitation secondary to AD; medications for nighttime management of insomnia or behavioral disturbances that included short-acting benzodiazepines, a low dose of alprazolam up to 0.5 milligrams (mg)/day, and a low dose of trazodone up to 50 mg/day; hypnotics for the treatment of insomnia; and certain classes of antidepressants.
Time Frame: up to Week 10
Population: mITT Population: all participants randomized in Stage 1 who had at least one post-Baseline NPI Agitation/Aggression score in Stage 1, and all placebo non-responders from Stage 1 who are re-randomized in Stage 2 and had at least one post-Week 4 NPI Agitation/Aggression score in Stage 2. Only those participants who took CMs were analyzed.
Measure: Number; unit: participants
Groups:
- AVP-923 in Stage 1/AVP-923 in Stage 2: Participants received oral AVP-923 during Stage 1 for 5 consecutive weeks. Participants received AVP-923-20 once daily (QD) in the morning and placebo in the evening (to maintain the blind) during the first week of Stage 1 (Days 1 to 7), AVP-923-20 twice a day (BID) during the next 2 consecutive weeks (Days 8 to 21), and AVP-923-30 BID the final 2 weeks of Stage 1 (Days 22 to 35). Participants who completed Stage 1 were eligible to participate in Stage 2 of the study. Participants continued to receive AVP-923-30 BID for the entire 5-week duration of Stage 2. Participants received AVP-923-20 QD in the morning and placebo in the evening (to maintain the blind) during the first week of Stage 2 (Days 36 to 42), AVP-923-20 BID during the next 2 consecutive weeks (Days 43 to 56), and AVP-923-30 BID the final 2 weeks of Stage 2 (Days 57 to 70).
- Placebo in Stage 1/AVP-923 in Stage 2: Participants receive matching oral placebo during Stage 1 for 5 consecutive weeks. Participants who completed Stage 1 were eligible to participate in Stage 2 of the study. Participants who were randomized to placebo in Stage 1 were stratified (based on their clinical response during Stage 1) into two subgroups (responders or non-responders) and were re-randomized to receive AVP-923 in Stage 2. Participants received AVP-923-20 QD in the morning and placebo in the evening (to maintain the blind) during the first week of Stage 2 (Days 36 to 42), AVP-923-20 BID during the next 2 consecutive weeks (Days 43 to 56), and AVP-923-30 BID the final 2 weeks of Stage 2 (Days 57 to 70).
- Placebo in Stage 1/Placebo in Stage 2: Participants receive matching oral placebo during Stage 1 for 5 consecutive weeks. Participants who completed Stage 1 were eligible to participate in Stage 2 of the study. Participants who were randomized to placebo in Stage 1 were stratified (based on their clinical response during Stage 1) into two subgroups (responders or non-responders) and were re-randomized to receive matching placebo BID throughout Stage 2.
Arm/Group | AVP-923 in Stage 1/AVP-923 in Stage 2 | Placebo in Stage 1/AVP-923 in Stage 2 | Placebo in Stage 1/Placebo in Stage 2
Number analyzed (Participants) | 84 | 53 | 58
participants
  Any change | 9 | 8 | 13
  Dose reduced | 1 | 0 | 1
  Dose increased | 0 | 1 | 1
  Change in frequency | 1 | 1 | 1
  Use discontinued | 2 | 2 | 2
  New usage | 7 | 6 | 11

22. Secondary Outcome: Number of Participants Using Rescue Medications
Description: Participants were allowed to receive oral lorazepam as rescue medication for the short-term treatment of symptoms of agitation, if deemed necessary by the investigator. Lorazepam was to be administered at doses up to 1.5 mg/day, and dosing was not to exceed 3 days in any 7-day period.
Time Frame: up to Week 10
Population: mITT Population
Measure: Number; unit: participants
Arm/Group | AVP-923 in Stage 1/AVP-923 in Stage 2 | Placebo in Stage 1/AVP-923 in Stage 2 | Placebo in Stage 1/Placebo in Stage 2
Number analyzed (Participants) | 93 | 59 | 66
participants
  Overall | 5 | 11 | 7
  Day 8 (Visit 2) | 0 | 3 | 1
  Day 22 (Visit 3) | 3 | 3 | 3
  Day 36 (Visit 4) | 5 | 3 | 3
  Day 43 (Visit 5) | 2 | 3 | 5
  Day 57 (Visit 6) | 1 | 3 | 4
  Day 70 (Visit 70) | 2 | 3 | 3

ADVERSE EVENTS:
Time Frame: up to Week 10
Description: Treatment-emergent adverse events (TEAEs), defined as AEs that first occurred, or worsened, after the first dose of study medication and within 30 days after the permanent discontinuation of the study medication (first dose date ≤ AE start date ≤ date of last dose + 30 days), are reported. TEAEs were collected in members of the Safety Population, comprised of all randomized participants who received at least one dose of study treatment.
Groups:
- AVP-923 in Stage 1/AVP-923 in Stage 2: Participants received oral AVP-923 during Stage 1 for 5 consecutive weeks. Participants received AVP-923-20 once daily (QD) in the morning and placebo in the evening (to maintain the blind) during the first week of Stage 1 (Days 1 to 7), AVP-923-20 twice a day (BID) during the next 2 consecutive weeks (Days 8 to 21), and AVP-923-30 BID during the final 2 weeks of Stage 1 (Days 22 to 35). Participants who completed Stage 1 were eligible to participate in Stage 2 of the study. Participants continued to receive AVP-923-30 BID for the entire 5-week duration of Stage 2. Participants received AVP-923-20 QD in the morning and placebo in the evening (to maintain the blind) during the first week of Stage 2 (Days 36 to 42), AVP-923-20 BID during the next 2 consecutive weeks (Days 43 to 56), and AVP-923-30 BID during the final 2 weeks of Stage 2 (Days 57 to 70).
Arm/Group | AVP-923 in Stage 1/AVP-923 in Stage 2 | Placebo in Stage 1/AVP-923 in Stage 2 | Placebo in Stage 1/Placebo in Stage 2
All-Cause Mortality (participants affected / at risk) | 0/93 | 0/59 | 0/68
Serious Adverse Events (participants affected / at risk) | 9/93 | 3/59 | 6/68
Other Adverse Events (participants affected / at risk) | 24/93 | 12/59 | 17/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AVP-923 in Stage 1/AVP-923 in Stage 2 (N=93) | Placebo in Stage 1/AVP-923 in Stage 2 (N=59) | Placebo in Stage 1/Placebo in Stage 2 (N=68)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Idiopathic Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 0 | 0 | 1
Acute Myocardial Infarction (Cardiac disorders) | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Chest Pain (General disorders) | 2 | 0 | 0
Kidney Infection (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Femur Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cerebrovascular Accident (Nervous system disorders) | 1 | 0 | 0
Transient Ischaemic Attack (Nervous system disorders) | 0 | 0 | 1
Aggression (Psychiatric disorders) | 0 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AVP-923 in Stage 1/AVP-923 in Stage 2 (N=93) | Placebo in Stage 1/AVP-923 in Stage 2 (N=59) | Placebo in Stage 1/Placebo in Stage 2 (N=68)
Diarrhoea (Gastrointestinal disorders) | 5 | 4 | 4
Urinary Tract Infection (Infections and infestations) | 5 | 3 | 4
Fall (Injury, poisoning and procedural complications) | 10 | 3 | 4
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1
Dizziness (Nervous system disorders) | 6 | 1 | 2
Agitation (Psychiatric disorders) | 3 | 1 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other